CLINICAL TRIAL: NCT02483117
Title: Adaptation and Validation of the Clinical Assessment Inventory (CIA) for Eating Disorders. Assessment of Its Relation With Other Clinical Measures
Brief Title: Adaptation and Validation of the Clinical Assessment Inventory for Eating Disorders (CIA)
Acronym: CIA
Status: Completed | Type: Observational
Sponsor: Hospital Galdakao-Usansolo (Other Government)
Collaborators: Carlos III Health Institute (Other Government)
Responsible Party: Principal Investigator, Josune Martin Corral, PhD, Hospital Galdakao-Usansolo
Other Study IDs: PS09/02012
Record Dates: First submitted 2015-06-17; First posted 2015-06-26 (Estimated); Last update posted 2015-06-26 (Estimated); Status verified 2015-06

CONDITIONS: Eating Disorders
MeSH Terms: conditions — Feeding and Eating Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Eating disorder patients by type of compensating behavior.: Data collection started in 2010; one year follow-ups were conducted through 2011-2012. Psychiatrists collaborating in the study informed personally their patients about the objectives of the study, and recorded the sociodemographic information, including age, gender, marital status, level of education, employment status, and people with whom the patient lived. Those who agreed to take part were also sent the questionnaires and informed consent form by mail. They were asked to return these by mail using an enclosed, pre-stamped envelope. Two reminders also were sent at intervals of 15 days to those who did not respond to the first mailing.
  Interventions: Other: Adaptation of the CIA

INTERVENTIONS:
Other: Adaptation of the CIA — Adaptation of the CIA into Spanish was performed using the backward-forward translation process, which ensures conceptual. Forward translation into Spanish was carried out by two independent native Spanish speaking translators who were fluent in English. Two other independent translators, totally blind to the original version, whose native language was English and who were fluent in Spanish, back-translated the consensus version into English. After reaching consensus on a final translated version, it was sent to the CIA's original author (Dr. Bohn) who gave her approval. We undertook a cognitive debriefing process with a group of 5 ED patients to identify any problems with language. The pre-final version was administered to two small groups, one made up of patients (a sample of 5 respondents) and the other of clinical experts (2 psychiatrists and 2 psychologists who were experts on ED).

SUMMARY:
The Clinical Impairment Assessment (CIA) assesses psychosocial impairment secondary to an eating disorder. The aim of this study was to create and validate a Spanish-language version of the CIA. Using a forward-backward translation methodology, we translated the CIA into Spanish and evaluated its psychometric characteristics in a clinical sample of 178 ED patients. Cronbach's alpha values, confirmatory factor analysis (CFA), and correlations between the CIA and the Eating Attitudes Test-12 and the Health-Related Quality of Life in ED-short form questionnaires evaluated the reliability, construct validity, and convergent validity, respectively. Known-groups validity was also studied comparing the CIA according to different groups; responsiveness was assessed by means of effect sizes.

ELIGIBILITY:
Inclusion Criteria:

* Outpatients were eligible for the study if they had been diagnosed with anorexia nervosa, bulimia nervosa, or an eating disorder not otherwise specified (EDNOS) by psychiatrists based on criteria established in the Diagnostic and Statistical Manual of Mental Disorders, 4th edition (DSM-IV) (American Psychiatric Association, 1994), and provided written informed consent to participate.

Exclusion Criteria:

* Patients were excluded if they had a malignant, severe organic disease, could not complete the questionnaires because of language barriers, or did not give written informed consent to participate in the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: We conducted a prospective study of all patients diagnosed with and treated for an ED in the Eating Disorders Outpatient Clinic of the Psychiatric Services at the Galdakao-Usansolo Hospital, in Bizkaia, Spain. This institution, which serves a population of 300,000 inhabitants, is part of the Basque Health Care Service, which provides free, unrestricted care to nearly 100% of the population. The diagnosis was verified via chart review. Throughout the 2-year study period, each patient received a psychopharmacologic and psychotherapeutic treatment program consisting of cognitive-behavioural treatment; nutritional orientation and counselling; psycho-education; motivational therapy; social skills training; and therapy to modify distorted perception of body image.
  Sample size was calculated according to the recommended 10:1 ratio of the number of subjects to the number of test items (Kline, 1998). The study was approved by the institutional review board of Galdakao-Usansolo Hospital.
Sampling Method: Probability Sample
Enrollment: 244 (Actual)
Dates: Start 2010-01; Primary Completion 2011-01 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
CIA questionnaire | Up to 2 years
  The CIA (v. 3.0) (Bohn et al., 2008) is a 16-item self-report measure of psychosocial impairment secondary to features of an eating disorder. This questionnaire measures three domains of impairment-personal, social, and cognitive-attributable to eating habits, exercising, or feelings about eating, shape, or weight over the previous 28 days. Items are rated on a four-point Likert scale, ranging from 0=''Not at all'' to 3=''A lot.'' A global CIA score ranging from 0 to 48 is calculated to provide a global index of the severity of psychosocial impairment due to eating disorder pathology during the past 28 days. A higher score indicates greater impairment. Subscale scores can be calculated to determine the three domains of impairment (personal, social, and cognitive). The original report of the CIA's psychometric properties supported adequate reliability and validity of the measure within a clinical sample of patients with eating disorders (Bohn et al., 2008).

SECONDARY OUTCOMES:
Eating Attitudes Test-12 (EAT-12) | Up to 2 years
  Eating problems were measured by the EAT-12 (Lavik, Clause & Pedersen, 1991). It uses a 4-point scale, from never (score 0) to always (score 2). The EAT-12 yields three factors: dieting, bulimia and food preoccupation, and oral control. Previous studies have supported its validity as a measure of disordered eating (Wichstrøm, Skogen & Øia, 1994; Wichstrøm, 1995). The internal consistency was a 0.71.
Health-Related Quality of Life in ED-short form (HeRQoLED-s) | Up to 2 years
  ED patients' quality of life was evaluated using the Health-Related Quality of Life in ED-short form (HeRQoLED-s) (Las Hayas et al, 2007; Las Hayas, Quintana, Padierna, Bilbao & Munoz, 2010). This questionnaire consists of 20 items distributed into two domains: social maladjustment and mental (α=0.91) and functional health (α=0.90). The higher the score, the lower the quality of life. This measure has been used successfully with Spanish-speaking populations (González, Padierna, Martín, Aguirre & Quintana, 2012; Las Hayas et al., 2006; Martín et al., 2011; Muñoz, 2009; Padierna et al., 2012).

CONTACTS AND LOCATIONS:
Overall Officials: Angel Padierna, MD, Principal Investigator — Hospital Galdakao-Usansolo

REFERENCES:
- [Result] Martin J, Padierna A, Unzurrunzaga A, Gonzalez N, Berjano B, Quintana JM. Adaptation and validation of the Spanish version of the Clinical Impairment Assessment Questionnaire. Appetite. 2015 Aug;91:20-7. doi: 10.1016/j.appet.2015.03.031. Epub 2015 Apr 1. PMID 25839732